CLINICAL TRIAL: NCT07194161
Title: Evaluation of the Impact of Pilonidal Cyst Recurrence on Quality of Life in Patients Previously Treated With Conventional Surgery or Laser Therapy
Acronym: SPIRIT
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-06-049-DARNIS-SPIRIT
Record Dates: First submitted 2025-09-12; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Pilonidal Cyst; Quality of Life
Keywords: pilonidal cyst; recurrence; quality of life; radical surgery; laser
MeSH Terms: conditions — Pilonidal Sinus; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- radical surgery
- laser treatment

SUMMARY:
The goal of this observational study is to describe the impact of recurrence on the quality of life of patients treated with radical surgery and laser therapy.

The secondary objective is to describe in patients treated with radical surgery and laser treatment :

* Intensity of pain and discomfort
* Duration of nursing care since surgery
* Duration of inactivity since intervention

DETAILED DESCRIPTION:
This is a single-centre exploratory study of patients previously treated for a pilonidal cyst who are consulting for a recurrence.

The study consists of a single assessment, the data from which will be recorded on an electronic case report form (CRF).

The objective of this study does not impose any particular constraints. The only evaluation of the study is carried out when the patient comes in for consultation for a recurrence of a pilonidal cyst.

Quality of life will be assessed using the The MOS 36-item short-form health survey (SF-36) scale and the Wound quality of life in Chronic Wounds survey (Wound QoL17).

Pain and discomfort will be assessed using a simple numerical scale ranging from 0 to 10.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 14 or over
* Patient has been informed of the objectives and conditions of the study and has not objected to the collection of his/her data.
* If the patient is under 18 years of age, both parents or the holder(s) of parental authority have been informed of their child's participation in the study and do not oppose it
* Presenting a recurrence of pilonidal sinus after a first complete treatment by radical surgery or laser

Recurrence is defined by :

* The presence of persistent troublesome symptoms more than 6 months after surgery: suppuration, iterative scar disunion, absence of healing despite care deemed optimal by the expert, recurrence of abscesses
* The presence of a characteristic MRI image, if this examination has been carried out: subcutaneous collection, in hyper T2.

Exclusion Criteria:

* Symptoms less than 6 months old
* First operation limited to simple abscess flattening
* Atypical symptoms, without radiological confirmation of recurrence: isolated pain, induration without inflammatory phenomena
* History of more than one elective surgery for pilonidal sinus
* Pilonidal sinus associated with a posteriorly developed anal fistula
* Persistence of a skin orifice, with no hair in it, without any symptoms
* Patient under court protection, guardianship or curatorship
* Mental deficiency or any other reason that may hinder comprehension of the information and non-opposition note0

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients consulting for a recurrence of pilonidal sinus previously treated as first-line treatment by radical surgery or laser.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Impact of recurrence of pilonidal cyst on patient's quality of life | Day 0
  Quality of life will be assessed using the SF36 scale. The SF-36 health status questionnaire has been validated in several languages, including English. It is a generic score for assessing quality of life. An average physical score (PCS = Physical Composite Score) and an average mental score (MCS = Mental Composite Score) can be calculated using an established algorithm. The SF-36 can be used by comparing (searching for correlations) the scores of the different domains of the SF-36 in a study population with those of the normal population, or by searching for correlations between the scores of the different domains of the SF-36 and other explanatory medical, functional, social, etc. variables.

SECONDARY OUTCOMES:
The intensity of pain and discomfort | Day 0
  The intensity of pain and discomfort will be assessed using a simple numerical scale ranging from 0 (no pain/discomfort) to 10 (worst pain/discomfort ever experienced).
Quality of life assessment with Wound QoL17 questionnaire | Day 0
  The Wound QoL17 is a questionnaire on quality of life in relation to chronic wounds. It comprises 17 items relating to the patient's experience over the last 7 days, which can be classified into three categories relating to daily life, the body and the psyche.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No